CLINICAL TRIAL: NCT00157092
Title: A Phase 1B/2A Study to Evaluate the Effect of Aerosolized, Recombinant Alpha 1-Antitrypsin on Epithelial Lining Fluid Analytes in Subjects With Alpha 1-Antitrypsin Deficiency
Brief Title: Study of the Effect of Aerosolized, Recombinant Alpha 1-Antitrypsin on Epithelial Lining Fluid Analytes in Subjects With Alpha 1-Antitrypsin Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Arriva Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 410302
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Alpha1-antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

INTERVENTIONS:
Drug: Aerosolized, Recombinant Alpha 1-Antitrypsin

SUMMARY:
The study was a Phase 1B/2A, uncontrolled, open-label, single-center study in individuals with congenital AAT (alpha 1-antitrypsin) deficiency. A baseline bronchoscopy with bronchoalveolar lavage (BAL) was performed 3 to a maximum of 4 weeks prior to the first administration of study drug. Fifteen eligible subjects were randomized to receive 1 of 3 dosing regimens of rAAT (100 mg daily, 100 mg twice daily, or 200 mg daily) administered via nebulization for 7 consecutive days. A post-treatment nadir BAL was obtained on study Day 8 (12 hours after last dose for subjects who receive drug therapy twice daily and 24 hours after the last dose for subjects who receive study product daily). BALs were conducted in the same lung lobe/segment. Follow-up visits took place on Day 15 and Day 36.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Male or female 18 years of age or older
* Documented, endogenous plasma AAT levels < 11 µM (< 80 mg/dL), either obtained from the medical history or, if not documented, plasma AAT measured after 28 day washout of any prior replacement therapy
* Forced expiratory volume at 1 second (FEV1) that is >= 50% of predicted, measured 30 minutes after a short-acting inhaled bronchodilator
* Arterial oxygen percent saturation (SaO2, measured using room air) within the normal limits for the individual study site
* For subjects receiving an inhaled corticosteroid, inhaled or oral β-2 agonist (e.g., albuterol via metered dose inhaler [MDI]) or inhaled anticholinergic bronchodilator (e.g., ipratropium bromide), or oral PDE (phosphodiesterase) inhibitor, treatment on a stable dose for at least 14 days prior to enrollment
* For any female of childbearing potential, a negative urine test for pregnancy within 3 days prior to enrollment and agreement to employ adequate birth control measures for the duration of the study
* No clinically significant abnormalities detected on a 12-lead electrocardiogram (ECG) performed at the screening visit
* Laboratory results obtained at the screening visit, meeting the following criteria:
* Serum aspartate transaminase (AST) and alanine transaminase (ALT) <= 2 times upper limit of normal range (ULN)
* Serum total bilirubin <= 2 times ULN
* < 2+ proteinuria on urine dipstick
* Serum creatinine <= 1.5 times ULN
* Absolute neutrophil count >= 1500 cells/mm3
* Hemoglobin >= 10.0 g/dL
* Platelet count >= 100,000/mm3

Exclusion Criteria:

* Clinically significant pulmonary impairment, other than emphysema and/or chronic bronchitis
* Moderate to severe bronchiectasis
* Clinically significant cardiac, hemostatic, or neurologic impairment, or other significant medical condition that, in the opinion of the investigator, would affect subject safety or compliance
* Psychiatric or cognitive disturbance or illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject safety or compliance
* Acute exacerbation of emphysema within 28 days prior to the screening visit
* Pregnancy or lactation
* Known history of allergy to yeast products
* Medical history precluding the use of epinephrine or other rescue medication for treatment of anaphylaxis
* Prior history of adverse reactions to the local anesthetic, sedative, BAL procedure, or pre-medication employed at the study center
* Use of oral or parenteral glucocorticosteroids, or alpha 1-antitrypsin replacement therapy within 28 days prior to baseline BAL, or any use planned during the study. However, the subject may enroll provided that a) consent is given to undergo a 28-day washout of the replacement or steroid therapy, and b) no study procedures are done until the washout is completed.
* Use of another investigational drug or investigational device within 28 days prior to baseline BAL
* Any upper or lower respiratory infection within 28 days prior to baseline BAL
* Having received a lung or liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-03-01 (Actual); Primary Completion 2004-10-14 (Actual); Study Completion 2004-10-14 (Actual)

PRIMARY OUTCOMES:
Alpha 1-antitrypsin levels assessed from epithelial lining fluid (ELF) samples | Baseline (minimum of 3 to a maximum of 4 weeks prior to the first administration of study product).
Alpha 1-antitrypsin levels assessed from epithelial lining fluid (ELF) samples | Day 8 after the first administration of study product

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States